CLINICAL TRIAL: NCT06937905
Title: A GCO Trial Exploring the Efficacy and Safety of Tarlatamab Versus Investigator-choice Chemotherapy in Pre-treated Patients With Advanced, Pulmonary or Gastroenteropancreatic Poorly Differentiated Neuroendocrine Carcinomas (NECs)
Brief Title: Tarlatamab vs Standard of Care Chemotherapy in Patients With Pre-treated Advanced, Pulmonary or Gastroenteropancreatic Poorly Differentiated Neuroendocrine Carcinomas (NECs)
Acronym: TARLANEC
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Intergroupe Francophone de Cancerologie Thoracique (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GCO-003
Record Dates: First submitted 2025-04-14; First posted 2025-04-22 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Neuroendocrine Carcinoma
Keywords: Neuroendocrine Carcinoma of Lung (Large cells); Gastroenteropancreatic Neuroendocrine Carcinoma; IFCT; FFCD; GERCOR; GCO
MeSH Terms: conditions — Carcinoma, Neuroendocrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A : Standard of care chemotherapy (Active Comparator): Study treatment in the arm A is left to the investigator appreciations. This may include immune checkpoint inhibitors, docetaxel, topotecan for primary lung tumors, and FOLFOX, FOLFIRI or alkylating-based chemotherapy in primary digestive tumors.
  Interventions: Drug: Standard of Care Chemotherapy
- Arm B : Tarlatamab (Experimental): Tarlatamab 10 mg every 2 weeks
  Interventions: Drug: Tarlatamab

INTERVENTIONS:
Drug: Standard of Care Chemotherapy — Study treatment in the arm A is left to the investigator appreciations. This may include immune checkpoint inhibitors, docetaxel, topotecan for primary lung tumors, and FOLFOX, FOLFIRI or alkylating-based chemotherapy in primary digestive tumors.
  Arms: Arm A : Standard of care chemotherapy
Drug: Tarlatamab — Tarlatamab 10 mg every 2 weeks
  Arms: Arm B : Tarlatamab

SUMMARY:
Based on the efficacy of tarlatamab in patients with small-cell lung cancer, we aim to assess the efficacy of tarlatamab in patients with Advanced, pulmonary (large-cell only) or gastroenteropancreatic neuroendocrine carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed consent:

   * Subjects must have signed and dated an IRB/IEC approved written informed consent form in accordance with regulatory and institutional guidelines. This must be obtained before the performance of any protocol related procedures that are not part of normal subject care.
   * Subjects must be willing and able to comply with scheduled visits, treatment schedule, and laboratory testing
2. Age ≥ 18 years.
3. WHO Performance status 0 - 1.
4. Life expectancy > 12 weeks.
5. Histologically proven and centrally confirmed poorly differentiated neuroendocrine carcinoma (NEC): large cells for lung NEC (WHO 2015 classification), and large and small cells for extra-gastroenteropancreatic (assessed on archived tissue, with possible pre-screening during first-line).
6. Expression of DLL3 in at least 1% of tumor cells (assessed on archived tissue, with possible pre-screening during first-line)
7. Tumor progression following one platinum based line of therapy.
8. Unresectable locally advanced or metastatic stage.
9. At least one measurable target lesion according to RECIST v1.1 per investigator assessment. The radiological assessment has to be done within the timelines indicated.
10. Adequate organ function: creatinine clearance > 50 mL/min, Neutrophils count ≥ 1500/mm3; Platelets > 100 000/mm3 ; Hemoglobin > 9 g/dL; AST and ALT < 3 x ULN (upper limit of normal) with total bilirubin ≤ 2 × ULN except subjects with documented Gilbert's syndrome or liver metastasis, who must have AST and ALT ≤ 5 x ULN and a baseline total bilirubin ≤ 3.0 mg/dL.
11. Full recovery from all toxicities associated with prior treatment, to acceptable baseline status, or a National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE v5.0) grade of 0 or 1, except for toxicities not considered a safety risk, such as alopecia or vitiligo.
12. Availability of tumor material for central review processes and translational research projects.
13. Absence of any unstable systemic disease and any psychological, familial, sociological or geographical factors potentially hampering compliance with the study protocol and follow-up schedule.
14. Females of childbearing potential who are sexually active with a non-sterilized male partner must use a highly effective method of contraception for 28 days prior to the first dose of investigational product, and must agree to continue using such precautions for 7 months after the final dose of investigational product; cessation of contraception after this point should be discussed with a responsible physician. Periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of contraception. They must also refrain from egg cell donation for 7 months after the final dose of investigational product.
15. Men who are sexually active with women of childbearing potential will be instructed to adhere to contraception for a period of 6 months after the last dose of treatment.
16. Patient covered by a national health insurance.

Exclusion Criteria:

1. Well-differentiated neuroendocrine tumor (NET G1, G2 and G3 according to digestive WHO 2017 classification or typical/atypical carcinoid tumor according to lung WHO 2015 classification)
2. Previous treatment targeting DLL3
3. More than one line of systemic therapy in the metastatic setting. Chemotherapy for non-metastatic stage is not considered as first-line if there is a time interval of at least 6 months between the last dose of chemotherapy for non-metastatic stage and the initiation of first-line chemotherapy for metastatic/recurrent disease.
4. Small cell lung NEC (except as a minor <30% component in mixed tumors)
5. Known EGFR activating mutation or ALK or ROS1 rearrangement for lung NEC
6. Untreated or symptomatic central nervous system (CNS) metastases:

   * Subjects with asymptomatic CNS metastases are eligible if clinically stable for at least 4 weeks and do not require intervention (including use of corticosteroids).
   * Subjects with treated brain metastases are eligible provided the following criteria are met:

     * Subject is asymptomatic from brain metastases
     * Whole brain radiation or surgery was completed at least 2 weeks prior to first dose of study treatment (stereotactic radiosurgery completed at least 7 days prior to first dose of study treatment)
     * Any CNS disease is clinically stable, subject is off steroids for CNS disease for at least 5 days (unless steroids are indicated for a reason unrelated to CNS disease), and subject is off or on stable doses of anti-epileptic drugs at least 14 days prior to first dose of study treatment
7. Leptomeningeal metastasis
8. Patients with a recent history of other malignancies except adequately treated non-melanoma skin cancer, and curatively treated in-situ cancer. Patients with history of solid tumors, including adenocarcinoma, treated in a curative way with or without chemotherapy and without any evidence of disease >2 years before randomisation can be included as well.
9. Major surgery within 28 days prior to initiation of study treatment.
10. Myocardial infarction and/or symptomatic congestive heart failure (New York Head Association class > class II) within 12 months prior to initiation of study treatment.
11. History of arterial thrombosis (e.g. stroke or transient ischemic attack) within 12 months prior to initiation of study treatment.
12. Symptoms and/or clinical and/or radiological signs suggestive of uncontrolled and/or acute active systemic infection within 7 days prior to first administration ofstudy treatment. Patient with active infection requiring parenteral antibiotic therapy. Upon completion of parental antibiotic therapy and resolution of symptoms, the patient may be considered eligible under the infection criterion.
13. Known sensitivity and/or immediate hypersensitivity to any component of study treatment.
14. History of primary immunodeficiency, history of organ transplant that requires therapeutic immunosuppression and the use of immunosuppressive agents within 28 days of randomization or a prior history of severe (grade 3 or 4) immune mediated toxicity from other immune therapy.
15. Patients with immune pneumonitis, pituitary or thyroid disorders, or pancreatitis under treatment with immuno-oncology agents.
16. Patients reporting infusion-related reactions or severe, life-threatening or recurrent immune-mediated adverse events (grade 2 or higher), including events leading to permanent discontinuation of immuno-oncology agents.
17. Presence of an indwelling line or drain (including the following: percutaneous nephrostomy tube, indwelling Foley catheter, biliary drain, peritoneal drain or catheter, pericardial drain or catheter, drain catheter or thoracic drain for pleural fluid collection).
18. Patient with a diagnosis of immunodeficiency or undergoing systemic corticotherapy or any other form of immunosuppressive therapy within 7 days prior to administration of the first dose of study treatment.
19. Known acute or chronic B or C hepatitis by serological evaluation. Patients with serological sequellae of hepatitis (antibodies test serologically positive for virus) without hepatitis could be included.
20. Known Human immunodeficiency virus infection
21. Patients who are pregnant or breast-feeding, or planning to become pregnant or breast-feed during the trial and within 7 months after the last dose of study treatment.
22. Male not wishing to abstain from sperm donation during the trial and within 6 months of the last study treatment.
23. Vaccination with live or attenuated virus vaccines is not permitted during the 28 days prior to administration of the first dose of treatment, and for the duration of the study. Vaccination against severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) should be avoided during selection, at least 14 days before the first day of treatment. Live, non-replicating smallpox vaccines (such as Jynneos) against monkeypox infection are permitted during the study (except during cycle 1) in accordance with the center's standard of care and internal recommendations.
24. Active autoimmune disease requiring systemic therapy (except replacement therapy) within the last 2 years or any other disease requiring immunosuppressive therapy during the study.
25. Patients with other concurrent severe and/or uncontrolled medical disease which could compromise participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Estimated)
Dates: Start 2026-02-06 (Actual); Primary Completion 2029-02-01 (Estimated); Study Completion 2030-08-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) in patients who received at least one dose of treatment. | About 4 years
  Time from date of inclusion to the date of death due to any cause.
  Time from date of inclusion to the date of death due to any cause.
  Time from date of inclusion to the date of death due to any cause.

SECONDARY OUTCOMES:
Safety and tolerability of cemiplimab | About 4 years
  Incidence, nature, and severity of treatment-related adverse events/treatment-emergent adverse events, graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events, Version 5.0 (NCI CTCAE v5.0)except CRS and ICANS events graded using ASTCT 2019
Objective Response Rate (ORR) | About 4 years
  Proportion of patients who have achieved a best overall response of complete response (CR) or partial response (PR) or stable disease (SD)
Duration of Response (DoR) | About 4 years
  Time from the date of the first response (CR or PR) to the earliest date of disease progression
Disease Control Rate (DCR) | About 4 years
  Proportion of patients who have achieved a best overall response of complete response (CR) or partial response (PR) or stable disease (SD)
Progression-Free Survival (PFS) | About 4 years
  Time from randomization to progression or death.
Overall survival (OS) | About 4 years
  Time from date of inclusion to the date of death due to any cause.
To evaluate the quality of life of patients with questionnaire EORTC Quality of Life Questionnaire - Core C30 (QLQ-C30) | About 4 years
  Time to symptom deterioration will be defined as the time from ranodmization until the date of first symptom deterioration.
  The European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire - Core Questionnaire C30 (EORTC QLQ-C30) is a 30 item instrument meant to assess some of the different aspects that define the quality of life of cancer patients.
  Scale : Not at all / A little / Quite a bit / Very much

CONTACTS AND LOCATIONS:
Locations (37):
- France (37):
  - Angers - CHU, Angers
  - Avignon - CH, Avignon
  - Besançon - CHU, Besançon
  - Boulogne - Ambroise Paré, Boulogne
  - Caen - CHU, Caen
  - Tours - CHU, Chambray-lès-Tours
  - Dijon - Centre Georges-François Leclerc, Dijon
  - Dijon - CHU Bocage, Dijon
  - Grenoble - CHU, Grenoble
  - Le Mans - CHG, Le Mans
  - Lille - Centre Oscar Lambret, Lille
  - Limoges - CHU, Limoges
  - Lyon - Centre Léon Bérard, Lyon
  - Lyon - Hôpital Edouard Herriot, Lyon
  - Lyon - Hôpital Privé Jean Mermoz, Lyon
  - Marseille - APHM, Marseille
  - Marseille - Institut Paoli-Calmettes, Marseille
  - Montpellier - CHU, Montpellier
  - Nice - Centre Antoine Lacassagne, Nice
  - Paris - Curie, Paris
  - Paris - Hôpital Cochin, Paris
  - Paris - Saint-Antoine, Paris
  - Paris - Tenon, Paris
  - Bordeaux - CHU, Pessac
  - Lyon - HCL, Pierre-Bénite
  - Poitiers - CHU, Poitiers
  - Reims - CHU, Reims
  - Rennes - CHU, Rennes
  - Rouen - CHU, Rouen
  - Nantes - Hôpital Laennec, Saint-Herblain
  - Nantes - Institut de Cancérologie de l'Ouest, Saint-Herblain
  - Strasbourg - Nouvel Hôpital Civil, Strasbourg
  - Toulon - CHI, Toulon
  - Toulouse - CHU, Toulouse
  - Tours - CHU, Tours
  - Vandoeuvre-lès-Nancy - Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy
  - Villefranche sur Saône - CH, Villefranche-sur-Saône

IPD SHARING:
Plan to Share IPD: Undecided